CLINICAL TRIAL: NCT05603975
Title: Analgesic Effect of Esketamine in Dressing Change for Severe Burns in Adults: a Prospective Randomized Controlled Study
Brief Title: Analgesic Effect of Esketamine in DCSB in Adultscontrolled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, ZhiHeng Liu, Director, Head of Anesthesiology, Principal Investigator, Clinical Professor, Shenzhen Second People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20223357006
Record Dates: First submitted 2022-10-20; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Analgesia; Burns
Keywords: Analgesia; Burn dressing change; Esketamine; Fentanyl; Adverse events
MeSH Terms: conditions — Agnosia; Burns | interventions — Esketamine; Injections, Intravenous; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was double-blind, including subjects, anesthesia operators, data collectors and dressing change operators. Nurse Song Yi opened the random envelope, diluted the drugs with normal saline according to the grouping information and filled them into a 10ml syringe. The syringe was labeled (marked with subject number, name and hospitalization number), and the grouping information was destroyed after confirmation, and confidentiality was strictly observed. Fully equipped drugs are given to the anesthesiologist and empty envelopes are given to the data collector.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EsKetamine Group (Active Comparator): The "Esketamine" was administered intravenously at 0.1mg per kilogram of body weight 1min before the dressing change.
  Esketamine Hydrochloride Injection 2ml：50mg
  Interventions: Drug: Esketamine 0.1mg/kg intravenous injection
- Control Group (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Esketamine 0.1mg/kg intravenous injection — The "Esketamine" was administered intravenously at 0.1mg per kilogram of body weight 1min before the dressing change.
  Arms: EsKetamine Group
Drug: Normal saline — The "Normal saline" was administered intravenously at 0.1ml per kilogram of body weight 1min before the dressing change.
  Other Names: Normal saline 0.1ml/kg intravenous injection
  Arms: Control Group

SUMMARY:
Patients with severe and above degree burns are often complicated with inhalation injury and systemic infection. During debridement and dressing change in such patients, doctors will be more cautious in using analgesics. Patients often moan, shiver and limb movement due to insufficient sedation and analgesia, resulting in unpleasant feelings and experiences, which increases the anxiety of patients during hospitalization. Previous studies have shown that the use of ketamine in burn patients during dressing change can produce good analgesia and maintain stable vital signs.

Esketamine, the dextral monomer of ketamine, has hypnotic, sedative and analgesic effects and could be safely used in clinical anesthesia. Compared with ketamine, esketamine has stronger analgesic efficacy and less circulatory influence, which is more consistent with the characteristics of ideal analgesic drugs in burn dressing. As an FDA-approved drug for the treatment of refractory depression, esketamine has potential social benefits in burn patients due to its rapid antidepressant pharmacological properties. This study hypothesized that esketamine could reduce the pain of dressing change in patients with severe burns and reduce the occurrence of early depression in such patients.

This study adopted a prospective, double-blind, randomized, controlled, single-center design. A total of 52 severe burn patients aged 18-60 years who need debridement and dressing change under sedation and analgesia were included and randomly divided into the experiment group: esketamine would be used in the induction phase; the control group: esketamine would not be used in the induction phase. Both groups were given dexmedetomidine and butofinol before induction, and fentanyl as a remedy during the dressing change phase. The dosage of fentanyl in the dressing change phase, the pain score (SF-MPQ) after recovery, the incidence of sedation-related complication were compared between the two groups.

This study explores the advantages of esketamine in reducing the use of opioids and the pain score of patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Grades II to IV
* Patients with severe degree burns Ages 18 to 60
* Patients who signed informed consent forms

Exclusion Criteria:

* Hepatic and renal insufficiency
* Allergy to intended medication
* History of antidepressant or antipsychotic drug use
* Atrioventricular block of second degree or higher
* Patients who can't cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The dosage of the remedy fentanyl | Within 5 minutes after the dressing change
  Observe the dose of syringe solution

SECONDARY OUTCOMES:
SF-MPQ score after awakening | Within 15 minutes to 30 minutes after the patient wakes up
  Evaluate Short-Form McGill Pain Questionnaire (SF-MPQ). The SF-MPQ is a highly reliable and sensitive instrument used to asses and measure pain levels. The minimum is 0 and the maximum is 60, with a higher score indicating more severe pain.
Incidence of sedation-related complication | From the beginning of the medication to the end of the dressing change, assessed up to 30 minute.
  The data collector observes and ticks the type of complication
Resuscitation time | From the end of the dressing change to the patient's Ramsay Sedation Scale was 1, assessed up to 10 minute.
  The data collector observed, filled in the end time of the dressing change and the time when the patient's Ramsay Sedation Scale was 1.
Incidence of early depression | 3 days after dressing change
  Evaluate Hospital Anxiety Depression
Incidence of nausea and vomiting | 1 days after dressing change
  Data collectors obtain data on the occurrence of events through patient or caregiver records
Proportion of patients taking fentanyl remedies | Within 5 minutes after the dressing change
  The proportion used is calculated from the data record
Patient satisfaction with dressing changes | 30 minutes to 1 hour after the patient wakes up
  Data collectors assessed patients using the VAS satisfaction score. The minimum is 0 and the maximum is 10, with a higher score indicating higher level of satisfaction.
Burn physician satisfaction with the procedure | Within 5 minutes after the end of the dressing change
  Data collectors assessed physician using the VAS satisfaction score. The minimum is 0 and the maximum is 10, with a higher score indicating higher level of satisfaction.
Incidence of serious complications associated with burns | 15 days after dressing change
  Collect data through electronic medical records

IPD SHARING:
Plan to Share IPD: No
The research protocol will be announced later in the plan.